CLINICAL TRIAL: NCT00050882
Title: A 12-Week Study Conducted at Multiple Centers, Blinded to Both the Patient and Doctor, Evaluating for Safety and Effectiveness Two Dosages of an Investigational Agent (GM-611) Versus a Placebo, That Are Randomly Assigned to Patients With Diabetic Gastroparesis
Brief Title: Safety and Effectiveness of an Investigational Agent (GM-611) in Patients With Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chugai Pharma USA (Industry)
Purpose: Treatment
Other Study IDs: GM-611-05
Record Dates: First submitted 2002-12-29; First posted 2002-12-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-02

CONDITIONS: Gastroparesis
Keywords: GM-611; Diabetic gastroparesis; Bloating; Delayed gastric emptying; Mitemcinal
MeSH Terms: conditions — Gastroparesis | interventions — mitemcinal

INTERVENTIONS:
Drug: GM-611

SUMMARY:
This study is intended to evaluate the potential to relieve the symptoms associated with gastroparesis during 12 weeks of treatment with oral tablets given twice a day of GM-611 5mg, 10mg or placebo to type I or II diabetics who require insulin.

Additionally the study will evaluate the safety and tolerability of GM-611 compared to placebo, the levels of GM-611 in the blood, and the possible effect of GM-611 on diabetic control.

ELIGIBILITY:
Inclusion Criteria:

Major Inclusion Criteria - Others Stipulated within the Protocol

The study physician must assure you have/are:

* Must be at least 18 years of age and have diabetes mellitus requiring insulin, which may be in addition to oral anti-diabetic agents.
* At least a three month history of the symptoms of gastroparesis that may include: early satiety (feeling full soon after beginning a meal), persistent fullness (long after eating), abdominal distention or bloating, nausea and vomiting. - No evidence of mechanical gastric obstruction, or other gastric problems since the onset of gastroparesis symptoms.
* You may be required to under go a Gastric Emptying Test (GET) procedure.
* You must be willing and able to maintain a daily telephone diary and consent to participate in this study.

Exclusion Criteria:

Major Exclusion Criteria - Others Stipulated within the Protocol

The study physician must assure you do not have/are not:

* Prior history of gastric surgery, excluding reflux surgery.
* Inability to withdraw from current prokinetic agents (e.g., metoclopramide, erythromycin, others) prior to, and during the study.
* Unstable current medical or surgical condition, or a recent history of frequent hospitalizations.
* A history of: HIV, recurring infection affecting the gastrointestinal track, cirrhosis, acute or chronic liver disease, active pancreatitis, cholecystitis, psychosis, severe depression, Parkinson's disease, myopathy, scleroderma, eating disorder, or organ transplant.
* Evidence or history of QT-prolongation, or use of drugs that are, or may be associated with QT-prolongation are prohibited.
* May not be pregnant, breast-feeding or not using approved methods of contraception.
* An allergy or intolerance to macrolide antibiotics (e.g., erythromycin).
* Use of any investigational drug within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - Arizona Center for Clinical Research, Glendale, Arizona
  - Lovelace Scientific Resources, Phoenix, Arizona
  - AGMG Clinical Research, Anaheim, California
  - Orange County Clinical Research, Inc, Cypress, California
  - Long Beach VA Medical Center, Long Beach, California
  - Research Foundation of America, Los Angeles, California
  - Community Clinical Trials, Orange, California
  - The Whittier Institute for Diabetes & Endocrinology, San Diego, California
  - Sharp Rees-Stealy Medical Group, San Diego, California
  - Westlake Medical Research, Westlake Village, California
  - Center for Diabetes & Endocrinology, Arvada, Colorado
  - Barbara Davis Center for Childhood Diabetes, Denver, Colorado
  - Gastroenterology Associates of Manatee, PA, Bradenton, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Anchor Research Center, Naples, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - BioQuan Research Group, North Miami, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Idaho Gastroenterology Associates, Boise, Idaho
  - Radiant Research Boise, Boise, Idaho
  - Rocky Mountain Institute of Clinical Research, Idaho Falls, Idaho
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Gastroenterology, Ltd., Peoria, Illinois
  - Rockford Gastroenterology Associates, Ltd, Rockford, Illinois
  - St. Vincent Hospital & Health Care Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Professional Research Network of Kansas, Wichita, Kansas
  - Digestive Health Center, University of Louisville, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Medical Research Institute, Slidell, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Center for Diabetes & Endocrinology, Grand Rapids, Michigan
  - Radiant Research, Edina, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - GI Associates Research, Jackson, Mississippi
  - University of Nebraska Health Center, Omaha, Nebraska
  - Lovelace Scientific Resources c/o Southwest Medical Associates, Las Vegas, Nevada
  - Core Health Services, Inc, Hampton, New Hampshire
  - Lovelace Scientific Resources, Inc, Albuquerque, New Mexico
  - Diabetic Care Associates, Binghamton, New York
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Prime Care Clinical Research, Clinton, Oklahoma
  - Regional Gastroenterology Associates of Lancaster, Lancaster, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University Hospital-GI Section, Philadelphia, Pennsylvania
  - Keystone Digestive Disorders Consultants, PC, Pittsburgh, Pennsylvania
  - Research Site, Stoneboro, Pennsylvania
  - Advanced Clinical Research, Ltd, North Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Diabetes Control Center, Orangeburg, South Carolina
  - Regional Research Institute, Jackson, Tennessee
  - Pharma Tex Research, Amarillo, Texas
  - Radiant Research-Dallas North, Dallas, Texas
  - Pro-Research Group, San Antonio, Texas
  - Diabetes & Glandular Disease Research Associates, San Antonio, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Metropolitan Research, Fairfax, Virginia
  - McGuire VA Medical Center, Richmond, Virginia
  - Evergreen Diabetes & Endocrinology Medical Group, Kirkland, Washington
  - Hyperion Clinical Research, Charleston, West Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin